CLINICAL TRIAL: NCT02470494
Title: The EarLens Contact Hearing Device (CHD) Spectrum Study
Acronym: Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EarLens Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP00009
Record Dates: First submitted 2015-06-08; First posted 2015-06-12 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sound amplificatoin via EarLens CHD (Experimental): Sound amplification provided via the EarLens CHD for subjects with hearing impairment.
  Interventions: Device: Sound amplification provided via the EarLens CHD

INTERVENTIONS:
Device: Sound amplification provided via the EarLens CHD — Subjects with mild to severe hearing impairment receiving sound amplification treatment with EarLens CHD.

SUMMARY:
The EarLens System is an assistive hearing device that is intended to provide amplification for the treatment of patients with sensorineural hearing impairment. The purpose of the proposed study (Extended Investigation under the Continued Access Policy) is to continue to allow access to the investigational medical device with the collection of device utility and clinic process-flow data while the marketing application is under review at the FDA.

DETAILED DESCRIPTION:
The study is designed to obtain observational data and as such no primary safety or efficacy endpoints or sample sizes are computed. Information gathered about device utility and clinic procedures from the physician, audiologist as well as subject questionnaires will be analyzed for the purpose of optimizing the process flow in different types of practice settings. A subset of relevant safety and efficacy measures from the Definitive Study (DEN150002) will be collected and adverse events will be tracked and reported per applicable regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years.
2. Mild to severe hearing impairment between 125 to 8000 Hz.
3. Asymptomatic of retro-cochlear lesions or cleared of retro-cochlear lesion by MRI.
4. No significant conductive hearing impairment;

   * No more than a 10 dB air-bone gap at 3 of 4 tested frequencies (500, 1000, 2000, or 4000 Hz)
   * Normal Type A tympanometry (indicating normal mobility of the tympanic membrane and middle ear bones)
5. Greater than or equal to 50% on clinical speech discrimination demonstrating an ability to benefit from amplification;
6. Able and willing to commit to the travel and time demands of the study (available for 5 months or longer) and able to comprehend and comply with the study materials and instructions
7. Experience with 1 or 2 air conduction hearing aids or previously evaluated for use with hearing aids;
8. Fluent speaker of American English due to use of American English study materials

Exclusion Criteria:

1. The Subject must not have known or active medical issues that would preclude having a hearing device, including:

   * an abnormal TM (deemed perforated, inflamed or has a dimeric or monomeric area, or in any other way abnormal);
   * an abnormal middle ear or a history of prior middle ear surgery other than tympanostomy tubes;
   * an ear canal anatomy that prevents the physician from seeing an adequate amount of the tympanic membrane.
   * an anatomical configuration of the external auditory canal that prevents satisfactory placement of the TMT
   * a history of chronic and recurrent ear infections in the past 24 months;
   * a rapidly progressive or fluctuating hearing impairment;
   * diagnosed with having a compromised immune system which may impact the tissue of the auricle or ear canal, such as keratosis obturans, ichthyosis, eczema of the auricle or ear canal, or received radiation of the head ever or chemotherapy for cancer within the last six years.
2. Must not fit the definition of a vulnerable subject, as per FDA regulations 21 CFR Parts 50 and 56

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Edwards, Study Director — EarLens, Corp.
Locations (8):
- United States (8):
  - California Hearing and Balance Center, La Jolla, California
  - Rodney Perkins Associates, Menlo Park, California
  - Camino Ear Nose and Throat Clinic, San Jose, California
  - University of Iowa, Iowa City, Iowa
  - CNC Hearing and Balance Center, Marrero, Louisiana
  - Carolina Ear and Hearing Clinic, Raleigh, North Carolina
  - Pittsburgh Ear Associates, Pittsburgh, Pennsylvania
  - Ear Medical Group, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arbogast TL, Moore BCJ, Puria S, Dundas D, Brimacombe J, Edwards B, Carr Levy S. Achieved Gain and Subjective Outcomes for a Wide-Bandwidth Contact Hearing Aid Fitted Using CAM2. Ear Hear. 2019 May/Jun;40(3):741-756. doi: 10.1097/AUD.0000000000000661. PMID 30300158

RESULTS

PARTICIPANT FLOW:
Groups:
- Sound Amplification Via EarLens CHD: Sound amplification provided via the EarLens CHD for subjects with hearing impairment.
  Sound amplification provided via the EarLens CHD: Subjects with mild to severe hearing impairment receiving sound amplification treatment with EarLens CHD.
Period: Overall Study
Arm/Group | Sound Amplification Via EarLens CHD
Started | 46
Completed | 41
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Sound Amplification Via EarLens CHD
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Hearing Stability Using Unaided Air Conduction Thresholds.
Description: Hearing sensitivity was monitored using earphones with the TMT (Tympanic Membrane Transducer) in place, but with the audio processor removed. Baseline and study end measurements were compared. A PTA4 (Pure Tone Average at 4 frequencies; 500, 1000, 2000 and 4000 Hz) was computed both for baseline unaided hearing post-placement with TMT in place, and unaided hearing with TMT in place at the 90-day for each ear, then averaged across both ears for each subject. A determination of "No Hearing Change" for the subject was made if the calculated hearing changes of the subject population are 10dB or less.
Time Frame: Baseline and up to 90-day.
Population: 40 subjects available for analysis between enrollment and 90-day measurement.
Measure: Mean (Standard Deviation); unit: dB difference in Unaided Hearing
Arm/Group | Sound Amplification Via EarLens CHD
Number analyzed (Participants) | 40
dB difference in Unaided Hearing | -0.5 (3.8)

2. Secondary Outcome: Change in Speech Understanding in Noise.
Description: The change in aided speech reception thresholds (SRTs) when compared to the baseline unaided condition was measured using a validated speech test, the HINT 90.
  Change in aided HINT 90 SRTs when compared to the baseline unaided condition. SRTs will be measured using HINT materials with the signal (speech level presented from 0 degrees) adapted relative to the noise (presented from 90 degrees held fixed at 60 dB SPL) to determine the signal-to-noise ratio for reporting the whole sentence correct 50% of the time (Nilsson et al., 1994). An improvement in HINT score is indicated as a negative (-) dB value change. A more negative value indicating an improvement of understanding speech and noise. An improvement of -1dB is equivalent to a 10% improvement in understanding speech and noise and is likely of clinical benefit. HINT 90 will be measured twice and averaged to obtain the per subject HINT SRT. All subject data will be averaged to obtain the means.
Time Frame: Baseline and up to 90-day.
Population: 28 subjects available for analysis between enrollment/treatment and 90-day measurement.
Measure: Mean (Standard Deviation); unit: dB difference in HINT scores
Arm/Group | Sound Amplification Via EarLens CHD
Number analyzed (Participants) | 28
dB difference in HINT scores | 2.0 (3.8)

3. Secondary Outcome: Change in Functional Gain Over the Frequency Range From 2000 to 10,000 Hz.
Description: 10 dB (decibel) change in the average pure tone thresholds for the subject population over the frequency range from 2000 to 10,000 Hz (2000, 3000, 4000, 6000, 8000, and 10,000 Hz). Measurement to be used in analysis are the baseline unaided soundfield (SF) thresholds measured prior to device placement and the aided soundfield thresholds measured 90-day post placement. Analysis includes calculation of the unaided soundfield thresholds minus aided soundfield thresholds
Time Frame: Baseline and up to 90-day.
Population: 40 subjects available for analysis between enrollment/treatment and 90-day measurement.
Measure: Mean (Standard Deviation); unit: dB difference in SF Hearing Thresholds
Arm/Group | Sound Amplification Via EarLens CHD
Number analyzed (Participants) | 40
dB difference in SF Hearing Thresholds | 27.2 (7.8)

4. Secondary Outcome: Change in Subject's Self-Perceived Ability to Communicate.
Description: The change in the subject's self-perceived ability to communicate with the use of the EarLens Device (CHD) when compared to baseline condition was measured using the validated Abbreviated Profile of Hearing Aid Benefit (APHAB) questionnaire. The APHAB produces scores for 4 subscales: Ease of Communication (EC), Reverberation (RV), Background Noise (BN), and Aversiveness (AV), which all range from 0-99%. A global score is computed by averaging the EC, RV, and BN subscores. For an individual score (either unaided alone or aided alone), a higher number indicates poorer performance, or more difficulty experienced. For this outcome measure, the difference between the average of the global unaided and aided scores is computed to determine the reduction (if any) in self-perceived difficulty, so a larger number in this outcome measure indicates better performance, as more of the difficulty has been reduced from the unaided condition by going to the aided condition.
Time Frame: Baseline and up to 90-day.
Population: 40 subjects available for analysis between enrollment/treatment and 90-day measurement.
Measure: Mean (Standard Deviation); unit: percentage of perceived benefit
Arm/Group | Sound Amplification Via EarLens CHD
Number analyzed (Participants) | 40
percentage of perceived benefit | 29.0 (17.1)

5. Other Pre Specified Outcome: Adverse Events
Description: All adverse events will be recorded on case report forms and determinations will be made as to the whether the events are Adverse Events, Serious Adverse Events, Unanticipated Adverse Device Effects and/or related to the investigational device or the procedure.
Time Frame: Baseline and up to 90-day.
Measure: Count of Participants; unit: Participants
Arm/Group | Sound Amplification Via EarLens CHD
Number analyzed (Participants) | 46
Participants
  Abrasion/blood/blister on tympanic membrane | 8
  Abrasion/blood/blister in ear canal | 34
  Ear discomfort/pain | 7
  Ear tip, other: swelling, itching | 1
  Inflammation/granulation tissue on TM | 3
  External otitis | 1
  TM perforation | 1
  Claustrophobia sensation | 1
  Other: Petechia and Erythemia | 2

ADVERSE EVENTS:
Time Frame: 90-days
Description: Subjects fitted with the Earlens Hearing Aid Device were evaluated for Adverse Events through 90-day follow-up.
Arm/Group | Sound Amplification Via EarLens CHD
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 34/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sound Amplification Via EarLens CHD (N=46)
Abrasion/blood/blister on tympanic membrane (Ear and labyrinth disorders) | 7 — Device and/or procedure related, anticipated, mild, all resolved.
Abrasion/blood/blister in ear canal (Ear and labyrinth disorders) | 25 — Device and/or procedure related, anticipated, mild/ moderate, all resolved.
Ear discomfort/pain (Ear and labyrinth disorders) | 5 — Device and/or procedure related, anticipated, mild/moderate, all resolved or improved.
Ear tip, other: swelling, itching (Ear and labyrinth disorders) | 1 — Device and/or procedure related, anticipated, mild, all resolved.
Inflammation/granulation tissue on TM (Ear and labyrinth disorders) | 3 — Device and/or procedure related, anticipated, mild, all resolved.
External otitis (Ear and labyrinth disorders) | 1 — Device and/or procedure related, anticipated, mild, all resolved.
TM perforation (Ear and labyrinth disorders) | 1 — Device and/or procedure related, anticipated, moderate, all resolved.
Claustrophobia sensation (Ear and labyrinth disorders) | 1 — Device and/or procedure related, anticipated, moderate, all resolved.
Other: Erythemia-pinpoint; or Petechia (Ear and labyrinth disorders) | 2 — Device and/or procedure related, anticipated, mild, all resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less